CLINICAL TRIAL: NCT02477150
Title: Immunogenicity and Safety of a Herpes Zoster Vaccine (Zostavax) in Patients With Systemic Lupus Erythematosus: a Randomized Controlled Trial
Brief Title: Safety and Immunogenicity of a Zoster Vaccine in SLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NTWC/CREC/15029
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLE (vaccine) (Active Comparator): Zostavax SC injection (0.65ml)
  Interventions: Biological: Zostavax
- SLE (placebo) (Placebo Comparator): Placebo SC injection (normal saline 0.65ml)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Zostavax — Vaccination of a zoster vaccine (Zostavax)
  Arms: SLE (vaccine)
Biological: placebo — placebo administration
  Arms: SLE (placebo)

SUMMARY:
To study the safety and immunogenicity of a herpes zoster vaccine in patients with SLE.

DETAILED DESCRIPTION:
Herpes zoster (HZ) (Shingles) is a painful condition caused by reactivation of varicella zoster virus (VZV) that remains dormant after primary infection. HZ reactivation may cause significant morbidity such as post-herpetic neuralgia and even mortality for disseminated infection, particularly in immunocompromised individuals.

HZ vaccine (Zostavax) is essentially a larger-than-normal dose of the chickenpox vaccine, which contains the Oka strain of live attenuated VZV. Zostavax has been shown to be safe and protective in immunocompetent elderly populations (>60 years of age) by reducing reactivation of HZ by 51% and post-herpetic neuralgia by 66%. Another study also demonstrated efficacy of Zostavax in reducing HZ infection by 70% in adults aged 50-59 years.

Data regarding the use of HZ vaccine in patients with rheumatic diseases are scant. A recent observational study involving 463,541 US patients with rheumatoid arthritis, inflammatory bowel disease, psoriatic arthritis and ankylosing spondylitis showed that 4% of patients had received HZ vaccination. After a median observation period of 2 years, the rate HZ reactivation among vaccinated patients was significantly lower than that of unvaccinated group (hazard ratio 0.61 [0.52-0.71]). Among 633 patients exposed to biologics at the time of vaccination, no cases of HZ or varicella infection occurred in the subsequent 42 days after vaccination. Thus, the vaccine appears to be safe in patients with autoimmune rheumatic diseases even receiving the biological agents.

HZ reactivation is fairly common in patients with systemic lupus erythematosus (SLE).

However, data regarding HZ vaccination in SLE patients are generally lacking. Safety and efficacy of HZ vaccination has recently been demonstrated in other immunocompromised groups such as HIV infection, post-chemotherapy and hematological malignancies. According to the 2011 EULAR recommendation, HZ vaccination may be considered in patients with autoimmune inflammatory rheumatic diseases provided that they are less seriously immunosuppressed.

The current study is designed to test for the immunogenicity and safety of a HZ vaccine (Zostavax) in patients with stable SLE who are receiving minimal immunosuppressive therapies for maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. SLE patients who fulfill ≥4 of the 1997 ACR (17) or the 2012 SLICC/ACR criteria for SLE (18)
2. Age ≥18 years
3. Clinically inactive disease with SELENA-SLEDAI score <6 (see below) and receiving stable dose of immunosuppressive agents for ≥6 months
4. History of varicella (chickenpox) or herpes zoster infection in the past
5. Willing to comply with all study procedures

Exclusion Criteria:

1. Active infection, including upper respiratory tract infection
2. Active untreated tuberculosis
3. Human immunodeficiency virus (HIV) infection
4. Lymphocyte count <500/mm2
5. Reduced serum IgG, IgA or IgM level (below normal range)
6. Serum creatinine >200umol/L
7. History of hematological malignancies (eg. lymphoma, leukaemia) and other solid tumors
8. Patients receiving doses of immunosuppressive agents exceeding the following:

   * Prednisolone (>15mg) or equivalent
   * Azathioprine (>100mg/day)
   * Mycophenolate mofetil (>1000mg/day)
   * Cyclosporin A (>100mg/day)
   * Tacrolimus (>3mg/day)
   * Methotrextate (>15mg/week)
   * Cyclophosphamide (any dose)
   * Biological agents eg. rituximab, belimumab (any dose)
9. Patients who are pregnant or plan to become pregnancy within one year of study entry
10. Patients who cannot give a written consent (mentally incapable or illiterate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
antibody rise to varicella zoster virus | 6 weeks
  Difference between the two groups in the proportion of patients who achieve a two-fold rise in IgG to VZV at week 6 post-vaccination compared to baseline

SECONDARY OUTCOMES:
safety (incidence of herpes zoster reactivation or chickenpox infection) | week 6
  incidence of herpes zoster reactivation or chickenpox infection
T cell response to VZV | week 6
  differences between IFN release upon VZV stimulation of PBMC

CONTACTS AND LOCATIONS:
Overall Officials: CC Mok, MD, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China

REFERENCES:
- [Derived] Mok CC, Chan KH, Ho LY, Fung YF, Fung WF, Woo PCY. Safety and immune response of a live-attenuated herpes zoster vaccine in patients with systemic lupus erythematosus: a randomised placebo-controlled trial. Ann Rheum Dis. 2019 Dec;78(12):1663-1668. doi: 10.1136/annrheumdis-2019-215925. Epub 2019 Sep 17. PMID 31530556